CLINICAL TRIAL: NCT05625815
Title: Evaluation of the Tolerance and Performance of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Brown Spots (Solar and Senile Lentigines, Post-inflammatory Hyperpigmentation)
Brief Title: Tolerance and Performance of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Brown Spots.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cryonove Pharma (Industry)
Collaborators: CEISO (Industry); Dermatech (Industry); Sefako Makgatho Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CS5_3
Record Dates: First submitted 2022-10-26; First posted 2022-11-23 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Solar Lentigo; Senile Lentigo; Post-inflammatory Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Condition 1: prototypes from (816-v1 001) to (816-v1 050) every day (Experimental): Application on the brown spots of the face and/or hands for the prototypes (816-v1001) to (816-v1 050) at D0, D1, D2, D3, D4 and D5.
  Interventions: Device: Prototypes (816-v1 001) to (816-v1 050)
- Condition 2: prototypes from (816-v1 051) to (816-v1 100) every week (Experimental): Application on the brown spots of the face and/or hands for the prototypes (816-v1 051) to (816-v1 100) at D0, D7, D14, D21, D28 and D35.
  Interventions: Device: Prototype (816-v1 051) to (816-v1 100)
- Conditions 3 : prototypes from (816-v1 101) to (816-v1 150) every two weeks (Experimental): Application on the brown spots of the face and/or hands for the prototypes (816-v1 101) to (816-v1 150) at D0, D14, D28, D42, D56 and D70.
  Interventions: Device: Prototypes (816-v1 101) to (816-v1 150)
- Condition 4 : prototypes from (816-v1 151) to (816-v1 200) every two weeks (Experimental): Application on the brown spots of the face and/or hands for the prototypes (816-v1 151) to (816-v1 200) at D0, D14, D28, D42, D56 and D70.
  Interventions: Device: Prototypes (816-v1 151) to (816-v1 200)

INTERVENTIONS:
Device: Prototypes (816-v1 001) to (816-v1 050) — Application on brown spots located on the face and/or the hand (6 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face or/and hand. Subjects will be lying supine, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 1: prototypes from (816-v1 001) to (816-v1 050) every day
Device: Prototype (816-v1 051) to (816-v1 100) — Application on brown spots located on the face and/or the hand (6 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face or/and hand. Subjects will be lying supine, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 2: prototypes from (816-v1 051) to (816-v1 100) every week
Device: Prototypes (816-v1 101) to (816-v1 150) — Application on brown spots located on the face and/or the hand (6 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face or/and hand. Subjects will be lying supine, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Conditions 3 : prototypes from (816-v1 101) to (816-v1 150) every two weeks
Device: Prototypes (816-v1 151) to (816-v1 200) — Application on brown spots located on the face and/or the hand (6 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face or/and hand. Subjects will be lying supine, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 4 : prototypes from (816-v1 151) to (816-v1 200) every two weeks

SUMMARY:
CS5_3 aims to evaluate the tolerance and to adjust the mode of administration of 4 different conditions of cryotherapy treatments applied on the brown spots of the face and hands with 3 prototypes. A brown spot is defined as solar or senile lentigo and post-inflammatory hyperpigmentation (PIH).

Each treatment corresponds to a combination of a specific sequence of a cryogenic spray and of a frequency of application.

The study will evaluate 3 prototypes :

* Prototype 1 : SN from (816-v1 001) to (816-v1 100)
* Prototype 2 : SN from (816-v1 101) to (816-v1 150)
* Prototype 3 : SN from (816-v1 151) to (816-v1 200)

Prototypes will be applied on the face and hands according to specific frequencies of application.

DETAILED DESCRIPTION:
Hyperpigmentation is a problem in all skin types. Safe depigmentation is a challenge. Cryotherapy with liquid nitrogen at -70 °C has been used in the treatment of solar skin lesions for many years but causes considerable damage.

Solar/senile lentigo is a harmless patch of darkened skin. It results from exposure to ultraviolet (UV) radiation, which causes local proliferation of melanocytes and accumulation of melanin within the skin cells (keratinocytes). Solar/senile lentigos or lentigines are very common, especially in people over the age of 40 years.

A solar/senile lentigo is a flat, well-circumscribed patch. It can be round, oval or irregular in shape. Colour varies from skin-coloured, tan to dark brown or black, and size varies from a few millimetres to several centimetres in diameter. They can be slightly scaly. Solar/senile lentigines are found as groups of similar lesions on sun-exposed sites, particularly the face or the back of hands.

Cryotherapy is more and more used to improve skin appearance and currently used to treat lentigo spot. However, the cryogenic gas (conventional cryotherapy - liquid nitrogen) creates a dermabrasion of the skin surface and person receiving this kind of treatment presents an impaired skin during a few days following the treatment as temporary damage of stratum corneum, erythema, scars, burns.

Following the side effects occurring after conventional cryotherapy application, the Sponsor has developed some devices using difluoroethane, manufactured by CRYONOVE PHARMA, already available on the local and international markets, e.g. CRYOBEAUTY MAINS and CRYOBEAUTY CORPS.

To continue its research and development activities, the sponsor has selected other sequences of a specific cryogenic spray (3 prototypes of devices for face and hands used according to different frequencies of application, i.e. 4 conditions evaluated) which has been used effectively and safely for lentigos treatment in Fitzpatrick phototypes I to IV on the face, with benefit for the subjects without any adverse safety outcomes. There is therefore a need to test the devices for lentigo and PIH on darker skin phototypes (V and VI according to Fitzpatrick scale), which also encounter hyperpigmentation challenges.

The rational for this study is to obtain a proof of performance on a representative panel sufficient to get statistically significant results of the expected effects. This will complete the data obtained during the previous proof of performance studies already performed on small panels as prerequisite data and have demonstrated an acceptable benefit/risk ratio.

Design:

The study is a proof of performance designed to be interventional, monocentric, randomized and double blinded.

Intervention:

Application on the skin of the face and the hands for the prototypes (816-v1 001) to (816-v1 200).

* Each spot will be treated by a defined prototype (always the same prototype on the same spot throughout the study) as given by a randomization list.
* Each spot will be treated 6 times during the study:

  * At D0, D1, D2, D3, D4 and D5) (condition 1)
  * At D0, D7, D14, D21, D28 and D35 (condition 2).
  * At D0, D14, D28, D42, D56 and D70 (conditions 3).
  * At D0, D14, D28, D42, D56 and D70 (conditions 4).

The distribution of the spots per phototypes and per condition is the following:

* Before any application, the dermatologist will collect the adverse events if any and will decide if the period between two consecutive applications should be extended or not.
* Before the application, the dermatologist will verify that the skin has not been treated by cosmetic products (no presence of cream that could interfere with the treatment) and is dry.
* Administration by the responsible technician (previously trained).
* Discontinuation of the treatment after the disappearance of the spot (to be confirmed by Dermatologist).
* Subjects will be lying supine, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down.
* During applications on the face, subjects will wear safety goggles protecting the eyes from cryogenic gas.
* From the start of the study until 2 months after the last treatment, volunteers will apply a sunscreen SPF 50+ (La Roche Posay, Anthelios if available to their hands and face in case of sun exposure). In case of prolonged sun exposure, application will be repeated as defined in the instructions for use.

ELIGIBILITY:
Inclusion Criteria:

* Female or male.
* Ages 18 to 75.
* Phototypes V and VI (according with Fitzpatrick scale), according to the spots distribution table.
* Featuring brown spots ≥ 3 and ≤ 6 mm in diameter on the face (and if possible, on the hands).
* Agreeing not to be exposed to the sun (or artificial UV) during the study.
* Informed, having undergone a general clinical examination attesting to his/her ability to participate in the study.
* Having given written consent for their participation in the study.
* No suspicion of carcinoma after investigation by a dermatologist.

Exclusion Criteria:

* Having performed cosmetic treatments (exfoliants, scrubs or self-tanners, manicures (only nails care acceptable), facials, UV ...) in the month before the start of the study, on the face and/or hands.
* Having applied a depilatory product in the month prior to the start of the study, on the face and/or hands.
* Having performed cosmetic treatments in a dermatologist (laser, intense pulse light, peeling, creams, cryotherapy ...), on the face and/or hands in the last 6 months.
* With dermatosis, autoimmune disease, systemic, chronic, or acute disease, or any other pathology that may interfere with treatment or influence the results of the study (people with diabetes or circulatory problems, allergic to cold, Raynaud's syndrome...).
* Receiving treatment by general or local (dermo corticoids, corticosteroids, diuretics ...) likely to interfere with the evaluation of the parameter studied.
* Participating in another study or being on a period of exclusion from a previous study.
* Unable to follow the requirements of the protocol.
* Vulnerable: whose ability or freedom to give or refuse consent is limited.
* Major protected by law (tutorship, curatorship, safeguarding justice...).
* People unable to read and write English language.
* Unable to be contacted urgently over the phone.

For female subjects:

* Pregnant woman (or wishing to be pregnant during study) or while breastfeeding.
* A woman who does not have a contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline skin hyperpigmentation | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70,Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots. A scale in 6 points (0 to 5) will be used :
  0=Clear of hyperpigmentation; 1= Almost clear of hyperpigmentation; 2=mild, but noticeable hyperpigmentation; 3=moderate hyperpigmentation (medium brown in quality); 4=severe hyperpigmentation (dark brown in quality); 5= very severe hyperpigmentation (very dark brown, almost black in quality).
Change from baseline skin hypopigmentation | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70,Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots. A scale in 5 points will be used (0 to 4): 0=no hypopigmented lesion; 1= very slight area of hypopigmentation of very small size and very slightly fairer than the surrounding skin; 2= slight area of hypopigmentation of small size and slightly fairer than the surrounding skin; 3= moderate : area of hypopigmentation of moderate size and much fairer than the surrounding skin; 4= severe : area of hypopigmentation of large size and much fairer than the surrounding skin.
Change from baseline skin appearance | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70,Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots and surrounded spotless skin area around the spot skin to assess erythema, oedema blister, bubble, scars, micro-bruise, hematoma, dryness,desquamation, fissures/cracks, roughness,crust, pink spots and papules. A scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe.
Change from baseline skin sensation | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70,Day 84 and Day 0 + 6 months
  The evaluation will be performed visually on the selected spots and around the spot skin to assess tightness, stinging, itching, warm and burning sensation. A scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe
Self-assesment of pain by the VAS | Day 0
  The pain of the treatment will be assessed by the Visual Analogue Scale (VAS) at time T0 on the treated area.
  The pain assessed is that felt during the application of the devices. It will be collected from the patient within 5 minutes of application. The VAS is made up of a 10-centimeter line anchored by two ends of the pain. One end is the "maximum pain imaginable". The other end is "no pain."
Change from baseline spots visibility | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70, Day 84, Day 0+6 months
  Standardized photographs will be taken using a Dermatoscope C-Cube® (PIXIENCE).The capture will be taken on the previously selected PIH/lentigo and a spotless area
Rating of spots and spotless areas visibility | Day 21, Day 49, Day 84
  Evaluation will be performed using a lentigines global improvement scale. Scoring of spots and spotless areas will be performed after the end of D84 visits on C-cube images by 3 dermatologists. It will be performed for each condition on pictures taken 2 weeks after the end of the treatment for the concerned condition.

SECONDARY OUTCOMES:
Self assessment of skin appearance | 0, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 70,Day 84 and Day 0 + 6 months
  The skin appearance will be assessed by subjects through a 3 items questionnaire with 5-point scale

CONTACTS AND LOCATIONS:
Locations (1):
- SMU - Photobiology Laboratory, Sefako Makgatho Health Sciences University, Pretoria, South Africa

IPD SHARING:
Plan to Share IPD: No